CLINICAL TRIAL: NCT06057090
Title: Do Certified Therapy Dogs Improve Behavior and Reduce Anxiety in Children Who Receive Administration of a Local Anesthetic for Dental Procedures? A Randomized Controlled Trial
Brief Title: Do Therapy Dogs Improve Behavior and Reduce Anxiety in Pediatric Dental Patients?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00129098
Record Dates: First submitted 2023-08-09; First posted 2023-09-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Therapy Animals; Dental Anxiety; Child Behavior; Anesthesia, Local
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy Dog (Experimental): This group will have a certified therapy dog present in the treatment room throughout the procedure. Prior to the procedure, the participant will be briefly introduced to the therapy dog and handler, who will remain in the room until the end of the procedure.
  Interventions: Behavioral: Therapy Dog
- Control (No Intervention): The control group receives standard of care and does not have a therapy dog present in the room during their treatment.

INTERVENTIONS:
Behavioral: Therapy Dog — Certified, volunteer therapy dogs and their handlers will be present in the room during procedures in the experimental arm to see if their presence reduces anxiety and improves behavior in pediatric dental patients.
  Arms: Therapy Dog

SUMMARY:
The goal of this clinical trial is to assess whether the presence of a certified therapy dog during dental procedures that require an injection reduces anxiety and improves behavior in pediatric dental patients.

The main questions it aims to answer are:

* Does the presence of a certified therapy dog during dental procedure requiring an injection reduce anxiety and improve behavior in pediatric dental patients?
* How do the parents of pediatric dental patients who participate in the study view the use of a certified therapy dog in their child's treatment?
* Does the presence of a certified therapy dog result in different concentrations of microbes in the treatment room?

All participants will receive standard of care. Researchers will compare the group with a therapy dog present to a group who does not have a therapy dog present to see if heart rate, oxygen saturation, percentage of nitrous oxide administered, and Frankl scores differ between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-7
* Children who are patients at the Medical University of South Carolina Department of Pediatric Dentistry
* Children classified as category 1 or 2 according to the American Society of Anesthesiologists Physical Status Classification
* Children whose parents/guardians are willing to consent to the child participating in the study
* Availability of parent to be present during treatment
* Children who require further care that includes the injection of a local anesthetic and whose procedure will take less than one hour

Exclusion Criteria:

* Patients whose cases are considered emergencies
* Patients who are classified as category 3 or higher according to the American Society of Anesthesiologists Physical Status Classification (6)
* If patient's medical status has worsened since initial evaluation
* Known allergy to dogs or other animals
* Past history of dental trauma
* Past history of animal bites or traumatic experience with a dog
* Emotional or developmental delays
* If, on the day of the treatment, patient presents with fever or other illness

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral measure, using the Frankl score | This behavior measure will be recorded at four timepoints: 1) immediately before the procedure, 2) during the procedure 3) during the procedure, and 4) immediately after the procedure
  Behavior will be recorded using the Frankl score, which ranges from 1 (definitely negative) to 4 (definitely positive)

SECONDARY OUTCOMES:
Parent survey responses | The surveys will be administered immediately after the procedure.
  Parents will be given a short survey about their child's participation in the study. Each arm of the study has its own survey. The survey for the control group is 4 multiple choice questions and one open-ended question. The survey for the experimental group contains 3 multiple choice questions and 1 open-ended question.
Microbial concentration | Experimental group: prior to arrival of therapy dog, and after departure of therapy dog. Control group: prior to arrival of participant, after departure of participant
  In the experimental arm, the dental operatory will be swabbed prior to the arrival of the therapy dog and again after the therapy dog as left. For the control group, the operatory will be swabbed.
Anxiety measure, heart rate | The heart rate will be recorded at four timepoints: 1) immediately before the procedure, 2) during the procedure 3) during the procedure, and 4) immediately after the procedure
  The participant's heart rate will be recorded, using a finger pulse oximeter
Anxiety measure, oxygen saturation | Oxygen saturation will be recorded at four timepoints: 1) immediately before the procedure, 2) during the procedure 3) during the procedure, and 4) immediately after the procedure
  The participant's oxygen saturation will be recorded, using a finger pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Marshall, PhD, Principal Investigator — James B. Edwards College of Dental Medicine, Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Pediatric Dental Clinic, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paryab M, Arab Z. The effect of Filmed modeling on the anxious and cooperative behavior of 4-6 years old children during dental treatment: A randomized clinical trial study. Dent Res J (Isfahan). 2014 Jul;11(4):502-7. doi: 10.4103/1735-3327.139426. PMID 25225565
- [Background] Vincent A, Easton S, Sterman J, Farkas K, Heima M. Acceptability and Demand of Therapy Dog Support Among Oral Health Care Providers and Caregivers of Pediatric Patients. Pediatr Dent. 2020 Jan 15;42(1):16-21. PMID 32075705
- [Background] Kamioka H, Okada S, Tsutani K, Park H, Okuizumi H, Handa S, Oshio T, Park SJ, Kitayuguchi J, Abe T, Honda T, Mutoh Y. Effectiveness of animal-assisted therapy: A systematic review of randomized controlled trials. Complement Ther Med. 2014 Apr;22(2):371-90. doi: 10.1016/j.ctim.2013.12.016. Epub 2014 Jan 6. PMID 24731910
- [Background] Casamassimo PS, Seale NS, Rutkauskas Ii JS, Rutkauskas JS. Are U.S. Dentists Adequately Trained to Care for Children? Pediatr Dent. 2018 Mar 15;40(2):93-97. PMID 29663907
- [Background] Stern J, Agarwal A, Pozun A. Pediatric Procedural Sedation. 2025 Mar 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK572100/ PMID 34283466
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509